CLINICAL TRIAL: NCT00004791
Title: Study of the Nutritional, Metabolic, and Body Composition Profile in Children and Adolescents With Epidermolysis Bullosa
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Baylor College of Medicine (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11912; BCM-H3246
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Epidermolysis Bullosa
Keywords: dermatologic disorders; epidermolysis bullosa; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Epidermolysis Bullosa; Skin Diseases; Genetic Diseases, Inborn; Rare Diseases

SUMMARY:
OBJECTIVES: I. Characterize the nutritional and metabolic profile of children and adolescents with epidermolysis bullosa.

II. Determine patterns of body composition in these patients. III. Determine the energy requirements of these patients by measuring resting energy expenditure.

IV. Assess protein nutrition by measuring lean body mass.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Data collected from a 5-day food diary are analyzed for protein, nutrient, and calorie intake. Nutritional, metabolic, and body composition are evaluated by indirect calorimetry, total body electrical conductivity, total body potassium, and lean body mass.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

* Epidermolysis bullosa
* Patient age: 2 months to 18 years

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15
Dates: Start 1995-08

CONTACTS AND LOCATIONS:
Overall Officials: William J. Klish, Study Chair — Baylor College of Medicine